CLINICAL TRIAL: NCT00975533
Title: A Randomized Study to Evaluate the Efficacy and Acceptability of Laparoscopic Placement of Gastric Modulator (TANTALUS® System) Versus Insulin Treatment in Obese Type 2 Diabetic Patients Sub-optimally Controlled With Oral Anti-diabetic Agents.
Brief Title: Gastric Modulator (TANTALUS® System) Versus Insulin Treatment in Obese Type 2 Diabetic Patients - a Randomized Control Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: MetaCure Limited (Industry)
Responsible Party: Simon Kin-Hung WONG, The Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2008.335
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2009-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tantalus (Experimental): The TANTALUS System is implanted using minimally invasive procedure (laparoscopy). It uses leads with stitch electrodes to deliver electrical signals to the gastric wall for the treatment of obese subjects with T2DM. The device is intended to improve glycemic control and induce weight loss.
  Interventions: Device: Tantalus
- Control (Active Comparator): Insulin treatment will be prescribed, in accordance with the common medical practice at the institute. Dosages will be recorded on a daily basis.
  Interventions: Drug: Insulin

INTERVENTIONS:
Device: Tantalus — The TANTALUS System is implanted using minimally invasive procedure (laparoscopy). It uses leads with stitch electrodes to deliver electrical signals to the gastric wall for the treatment of obese subjects with T2DM.
  Arms: Tantalus
Drug: Insulin — Insulin treatment will be prescribed, in accordance with the common medical practice at the institute. Dosages will be recorded on a daily basis.
  Arms: Control

SUMMARY:
This study aims to analyze the pre- and post-operative clinical, hormonal and biochemical changes in moderately obese type 2 diabetic patients who are sub-optimally controlled on at least 2 anti-diabetic agents. Study participants will either receive implantation of the gastric contraction modulator or conventional treatment with insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Adult patients aged between 18 and 60 years (inclusive)
* Male or female of Chinese ethnicity
* Type 2 diabetes mellitus with disease duration of greater than 2 and less than 10 years
* severe obesity, includes BMI 25 to 27.5 kg/m and central obesity defined by waist circumference greater than 90 cm in women and greater than 95 in men, or BMI greater than 27.5 to less than 35 kg/m
* HbA1c greater than or equals to 7.5% but less than 10% despite treated with maximum dose or maximally tolerated dose of 2 anti-diabetic drugs (OAD) with good drug compliance

Exclusion Criteria:

* On anti-obesity drugs
* On insulin treatment at the time of the recruitment
* On glitazone or incretins (dipeptidyl peptidase-4 inhibitor or glucagons-like peptide-1) treatment
* On any implantable device including cardiac pacing
* Anticipated to have MRI examinations
* Fasting C-peptide level less than 0.5g/L
* Renal impairment (defined as serum creatinine greater than 150mol/L and/or estimated glomerular filtration rate less than 60 mL/min/1.73m)
* Significant liver impairment (ALT more than 3 times upper limit of normal range)
* Active malignant disease. Patients with malignant disease who have been disease-free for at least 5 years are eligible
* Active infection
* Active and uncontrolled thyroid diseases
* Childbearing age female patients without reliable contraceptive methods
* Life expectancy less than 12 months
* Administration of another investigational drugs or procedures within 4 weeks before screening
* Any medical illness or condition as judged by the investigators as ineligible to participate the study
* Special population, e.g. prisoner, mentally disabled, investigators' student or employees

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-07 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
changes in body weight before and after interventions at 6 and 12 months | 6 months and 1 year
changes in HbA1c before and after interventions | 6 and 12 months
frequency of hypoglycaemia | 6 month and 1 year
dichotomous composite end point assessing the proportion of patients meeting all of the following prespecified criteria defined as: 1. HbA1c ≤7.0% or an HbA1c reduction from baseline ≥0.5% 2. no weight gain 3. no severe hypoglycaemia | 6 and 12 months
composite quantitative score calculate from the results of glycemic control, weight response and degree of hypoglycemia | 6 month and 1 year

SECONDARY OUTCOMES:
waist circumferences | 6 month and 1 year
insulin secretory responses (as measured by the standard meal test) | 6 month and 1 year
Hormonal profiles (including gut hormones) | 6 months and 1 year
a. eating behavior, satiety and quality of life as measured by the Food Frequency Questionnaire, Visual Analogue Rating Scale To Assess Satiety, EDE, SF-36 and GIQOL questionnaires | 6 month and 1 year
resting energy expenditure as monitored by indirect calorimetry (MedGem). | 6 month and 1 year
radiological assessment (ultrasound scan and densitometry to measure mesenteric and total body fat respectively) | 6 months and 1 year
differences in insulin requirement | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Simon KH Wong, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong, China

REFERENCES:
- [Derived] Wong SK, Kong AP, Luk AO, Ozaki R, Ng VW, Lebovitz HE, Ng EK, Chan JC. A pilot study to compare meal-triggered gastric electrical stimulation and insulin treatment in Chinese obese type 2 diabetes. Diabetes Technol Ther. 2015 Apr;17(4):283-90. doi: 10.1089/dia.2014.0234. Epub 2015 Feb 24. PMID 25710812